CLINICAL TRIAL: NCT00330629
Title: Preference and Vegetarian Diet in Weight Loss Treatment
Acronym: PREFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lora Burke, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000674; R01DK058631 (NIH)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Behavioral Treatment (Active Comparator): Goal setting: daily/weekly goals for calorie and fat consumption, exercise time, and behavior change.
  Self-monitoring: systematically observing and recording one's behavior,45,46 which will be reviewed by the therapists, and written feedback will be provided to reinforce positive behaviors.
  Feedback: therapists monitor the recorded behavior changes and provide feedback/encouragement.
  Interventions: Behavioral: Standard Behavioral Treatment
- SBT+LOV Group (Active Comparator): In addition to SBT, participants will aim to eliminate all meat, poultry, and fish from their diet over the first 6 weeks, and will be taught how to select appropriate substitutes for these foods, such as low- or no-fat dairy products (cheeses, milk), and protein-containing vegetable sources (soy products, legumes). .
  Interventions: Behavioral: Standard Behavioral Treatment; Behavioral: SBT+LOV

INTERVENTIONS:
Behavioral: Standard Behavioral Treatment — Participants in this condition will receive the standard behavioral treatment (SBT) described above. Food tastings will be held at the sessions and will focus on fat modified food products.
Behavioral: SBT+LOV — The focus will be on the elimination of meat products as a means to reduce fat intake.
  Arms: SBT+LOV Group

SUMMARY:
We propose to add a treatment preference component to a larger study testing standard behavioral treatment (SBT) for weight loss without specific food group restriction vs standard behavioral treatment with gradual elimination of meat, poultry, and fish [a lacto-ovo-vegetarian (LOV) meal plan]. Eligible respondents will be randomized to one of two conditions: Treatment Preference-Yes/No. Individuals in the Treatment Preference-Yes will be assigned to their choice (SBT or SBT+LOV), those in Treatment Preference-No will be randomized to either SBT or SBT+LOV without regard to their preference.

DETAILED DESCRIPTION:
Both groups will receive the behavioral treatment program (32 sessions over 12 months) that has been used successfully in numerous behavioral weight loss studies conducted by Dr. Wing.42-44 The Treatment Preference-Yes and -No Groups will meet on separate evenings to avoid contamination across the conditions but will be led by the same multidisciplinary team (behavioral scientists, nutritionist, exercise physiologist). A brief description of elements common to both groups follows:

Group Sessions: Groups will meet for 45-60 minutes weekly for Months 1-6, bi-weekly for Months 7-9, and monthly for Months 10-12. Participants will be weighed, receive nutritional and behavioral counseling, turn in the weekly diaries, and receive homework assignments at the sessions.

Dietary Restrictions: Calorie Goal. Participants will receive an individualized calorie goal calculated from baseline body weight (1200 calories < 200 lbs; 1500 calories for > 200 lbs), used successfully in previous studies.42 Fat Goal. Fat gram goals will approximate 25% of calories.

Physical Activity and Exercise: Participants will gradually increase their exercise, primarily walking, until they reach a minimum goal of 150 minutes per week (a caloric expenditure of 1000 calories/wk).

Behavioral Strategies to Use in Changing Eating and Exercise Habits: The central features follow:

Goal setting: daily/weekly goals for calorie and fat consumption, exercise time, and behavior change.

Self-monitoring: systematically observing and recording one's behavior,45,46 which will be reviewed by the therapists, and written feedback will be provided to reinforce positive behaviors.

Stimulus control: behavioral strategies designed to assist participants in altering their environment, minimize the cues that might trigger problematic behaviors, and add cues to increase activity.10 Problem solving: consists of 5 steps: identifying the problem; brainstorming solutions; evaluating the pros/cons of each potential solution; implementing the solution plan; and evaluating its success.47,48 Social assertion: use assertive skills in situations that may threaten their meeting eating/exercise goals.

Feedback: therapists monitor the recorded behavior changes and provide feedback/encouragement.

Cognitive strategies: taught how to recognize patterns of negative thought that can interfere with behavior change, how to counter these negative thoughts, and to use positive self-statements.

Relapse prevention: recognize situations that place them at risk for lapses49 Maintenance: weight loss maintenance will be addressed, identify their own problems related to maintaining their new patterns of eating/exercising, develop problem-solving strategies.50-53 Reinforcement: provide a magazine subscription to reinforce what is learned in each group.

Ensuring dietary adequacy: diaries will be reviewed weekly for energy intake and expenditure and for nutrient adequacy. A dietitian will be part of the team reviewing the diaries.

Incentives: will be given a monetary incentive for completing the paper-and-pencil instruments, Three-Day Food Record, and appointment for phlebotomy at 6, 12, and 18 months, and for completing the Final Visit.

Educational Session on Risk of Cholelithiasis: A brief (~15-20 minutes with Questions and Answers to follow) educational session will be provided to study participants informing them of risk factors for cholelithiasis. The information presented will include predisposing risk factors (i.e., overweight/obesity at baseline, rapid weight loss, inadequate calorie and fat gram intake) and guidelines for reducing risk for cholelithiasis (i.e., safe rate of weekly weight loss, minimal caloric and fat gram intake per day). Participants will also be provided with an informational letter on cholelithisis risk factors and risk reduction and will be asked to sign this letter and return it to the staff on the project, to be placed in their study participant files.

c.6.2. Dietary Intervention The treatment conditions will differ in eating plans and breadth of content (e.g., cooking classes, grocery shopping field trips) to better assist and support SBT+LOV participants develop their skills to implement and maintain the vegetarian meal plan. The differences are described below.

c.6.2.1. Group 1: Dietary Intervention for the Standard Behavioral Treatment Group Participants in this condition will receive the standard behavioral treatment (SBT) described above. Food tastings will be held at the sessions and will focus on fat modified food products.

c.6.2.2. Group 2: Dietary Intervention for the SBT+LOV Group Diet: In addition to SBT, participants will aim to eliminate all meat, poultry, and fish from their diet over the first 6 weeks, and will be taught how to select appropriate substitutes for these foods, such as low- or no-fat dairy products (cheeses, milk), and protein-containing vegetable sources (soy products, legumes). The focus will be on the elimination of meat products as a means to reduce fat intake.

Self-monitoring: In addition to energy intake/expenditure, record the number of meat meals eaten.

Social support for dietary changes: One session will be offered: an overview of the eating pattern, how to merge different eating styles in one family, how to dine at the same restaurant, and how to attend family and social functions. Participants will be encouraged to bring family members. Family members will not be considered as subjects in the study and will not be asked to provide any information. They will be there as guests to receive information that may allow them to better support their family member who is participating in the study.

Modeling: Practicing vegetarians will share strategies on making the transition to a vegetarian diet.

Ensuring dietary adequacy: Menstruating females will be instructed to use vegetarian sources of iron (e.g., legumes, dark leafy greens, dried fruits) and to use iron supplements if their iron intake does not appear adequate on their reported diet. Hemoglobin will be measured at each assessment point and results will be reported to patient's physician if value is below normal. The cost for this test will be covered by the grant.

ELIGIBILITY:
Inclusion Criteria:

* (1) be 18 to 55 years of age; (2) have a BMI of at least 27 but not greater than 43; (3) be willing to be randomized to one of the two preference conditions (Yes/No) and one of the two treatment conditions (SBT or SBT+LOV); and (4) have successfully completed a 5-day diary

Exclusion Criteria:

* (1) presence of a current serious illness or unstable condition (e.g., acute myocardial infarction or diabetes) for which physician supervision of diet and exercise prescription is needed; (2) presence of cardiovascular or orthopedic condition that would require physician clearance prior to participation; (3) limitations precluding ability to exercise; (4) pregnancy or intention to become pregnant in the next 18 months; (5) current treatment for a psychological disorder; (6) reported alcohol intake >4 drinks/day; (7) current or recent (past 6 months) participation in a weight loss treatment program or use of weight loss medication; (8) reporting no regular intake of meat, fish, and fowl; or presence of a serious binge eating problem

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2002-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
weight change at 18 months | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lora E. Burke, PhD, MPH, RN, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Goode RW, Ye L, Sereika SM, Zheng Y, Mattos M, Acharya SD, Ewing LJ, Danford C, Hu L, Imes CC, Chasens E, Osier N, Mancino J, Burke LE. Socio-demographic, anthropometric, and psychosocial predictors of attrition across behavioral weight-loss trials. Eat Behav. 2016 Jan;20:27-33. doi: 10.1016/j.eatbeh.2015.11.009. Epub 2015 Nov 14. PMID 26609668
- [Derived] Warziski MT, Sereika SM, Styn MA, Music E, Burke LE. Changes in self-efficacy and dietary adherence: the impact on weight loss in the PREFER study. J Behav Med. 2008 Feb;31(1):81-92. doi: 10.1007/s10865-007-9135-2. Epub 2007 Oct 26. PMID 17963038
- [Derived] Burke LE, Hudson AG, Warziski MT, Styn MA, Music E, Elci OU, Sereika SM. Effects of a vegetarian diet and treatment preference on biochemical and dietary variables in overweight and obese adults: a randomized clinical trial. Am J Clin Nutr. 2007 Sep;86(3):588-96. doi: 10.1093/ajcn/86.3.588. PMID 17823421